CLINICAL TRIAL: NCT01470001
Title: The Effect of Solifenacin on Post Void Dribbling in Women: A Randomized Controlled Multicenter Trial
Brief Title: The Effect of Solifenacin on Post Void Dribbling in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0513
Record Dates: First submitted 2011-11-02; First posted 2011-11-10 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Post-micturition Incontinence; Incontinence
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- solifenacin (Active Comparator): patients in this arm will receive drug
  Interventions: Drug: solifenacin
- placebo (Placebo Comparator): patients is this arm will receive placebo
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: solifenacin — patient will receive solifenacin 5mg daily or placebo daily
  Other Names: vesicare

SUMMARY:
This is a double-blind, randomized, controlled, parallel design (n=140) study with the purpose of measuring the efficacy of Solifenacin 5mg in the treatment of women with Post Void Dribbling.

DETAILED DESCRIPTION:
This investigation will have a double-blind, randomized, and controlled, parallel design with the % reduction in post void dribbling episodes (events) as the primary endpoint.

Secondary endpoints will include:

1. The % of patients with at least a 50% reduction in post void dribbling episodes.
2. Patient's perspective of the impact of their disease, which will be captured using the Pelvic Floor Distress Inventory, and another questionnaire that asks about urinary symptoms and quality of life.

We will compare Solifenacin 5 mg to placebo. 140 subjects will be enrolled, with 70 subjects in each arm. The treatment group will receive 5mg of Solifenacin daily for 12 weeks. Astellas Pharma will be supplying both drug and placebo, they will be prepackaged and numbered. The Pharmaceutical Research Center will randomly assign subjects into the treatment vs. placebo group blinding both the subjects and investigators

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 18 and 89
2. Incontinence in the form of post void dribbling that occurs at least twice weekly.

Exclusion Criteria:

1. Severe renal or hepatic disease.
2. Active urinary tract infection.
3. Glaucoma.
4. Stress incontinence as the only incontinence symptom
5. Urge incontinence as the only incontinence symptom
6. Chronic severe constipation.
7. History of bladder cancer.
8. Known or suspected hypersensitivity to anticholinergics.
9. Any clinical condition that would not allow safe completion of the study.
10. Pregnancy or lactation, intention to become pregnant during the study, or use of an unreliable birth control method in women of childbearing potential. Reliable forms of contraception include: permanent sterilization of either partner, hormonal contraception (oral contraceptive, Nuva ring, contraceptive patch, depoprovera, implants), intrauterine device (IUD), and condoms. Abstinence is considered a reliable form of contraception, but abstinent subjects will be informed that they need to use condoms or other form of birth control mentioned above if they become sexually active during the study.
11. Presently on systemic anti-cholinergic therapy or who have been on therapy within the last 4 weeks. Anti-cholinergic drugs include; darifenacin, fesoterodine, hyoscyamine, oxybutynin, solifenacin, tolterodine, and trospium.
12. Solid forms of potassium supplementation, as this presents an increased risk of GI side effects.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tova S Ablove, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: study subjects who received solifenacin 5mg daily
- Placebo: study subjects who received placebo daily
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 58 | 60
Completed | 53 | 58
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin | Placebo | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (14.2) | 48.2 (12.8) | 51.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 56 | 59 | 115
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 51 | 52 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 58 | 60 | 118
post void dribbling episodes per day [Mean (Standard Deviation); unit: post void dribbling episodes] | 3.38 (2.84) | 3.11 (2.65) | 3.25 (2.76)
voids per day [Mean (Standard Deviation); unit: voids per day] | 9.55 (5.20) | 9.23 (3.68) | 9.39 (4.48)
urgency episodes per day [Mean (Standard Deviation); unit: urgency episodes per day] | 2.64 (2.84) | 2.87 (4.73) | 2.76 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: The Percent Reduction in Post Void Dribbling Episodes (Events)
Time Frame: outcome measures will be assessed at week 0 (baseline), and compared to an average measure of weeks 10 through 12
Population: one subject was excluded from analysis because of missing baseline data
Measure: Mean (Full Range); unit: percent reduction
Arm/Group | Solifenacin | Placebo
Number analyzed (Participants) | 58 | 59
percent reduction | 59.8 [44.0 to 75.7] | 42.1 [26.8 to 57.4]
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; A planned sample size of 56 subjects per group provided 80% power to detect a difference of 0.25 between post void dribbling response rates (assumed to be 0.35 under the null hypothesis and 0.60 under the alternative hypothesis) at a one-sided 0.05 significance level; Test type: Superiority or Other; p = .1135, Mixed Models Analysis; mixed model with repeated measurements; Mean Difference (Final Values) = 17.7, 95% CI 2-sided [-4.3 to 39.7]

2. Secondary Outcome: the Percent of Patients With at Least 50% Reduction in Post Void Dribbling Episodes
Time Frame: outcome measures will be assessed at week 0 (baseline), and compared to an average measure of weeks 10 through 12
Population: one study subject was excluded form analysis due to missing baseline data
Measure: Number; unit: percent
Arm/Group | Solifenacin | Placebo
Number analyzed (Participants) | 58 | 59
percent | 69.8 | 55.5
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; Test type: Superiority or Other; p = .0919, Regression, Logistic; logistic regression with repeated measurements; Mean Difference (Net) = 14.3, 95% CI 2-sided [-2.3 to 30.8]

3. Secondary Outcome: Change in Patients Perspective of the Impact of Their Disease, Captured Using the Pelvic Floor Distress Inventory (Urinary Questions)
Description: The difference between baseline and follow up (last 20 days on drug) scores was the recorded measure. The larger the negative # the greater the effect.
  The survey was divided into 3 sections, each section worth 100 points. Total scores could range from 0 to 300 (0 no disease, 300 severe disease).
Time Frame: outcome measures will be assessed at week 0 (baseline), and compared to an average measure of the last 20 days on placebo or treatment
Population: one subject was excluded from analysis because of missing baseline data
Measure: Mean (Full Range); unit: change in score
Arm/Group | Solifenacin | Placebo
Number analyzed (Participants) | 58 | 59
change in score | -35.12 [-130 to 32.57] | -28.84 [-130 to 65.15]
Statistical Analysis 1: Comparison: Solifenacin vs Placebo; the difference in change between the groups was measured; Test type: Superiority or Other; p = 0.44, ANCOVA — p value was adjusted for age; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-17.5 to 6.2] — we calculated the estimated difference in change between the placebo and treatment groups

ADVERSE EVENTS:
Arm/Group | Solifenacin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/58 | 0/60
Other Adverse Events (participants affected / at risk) | 23/58 | 16/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin (N=58) | Placebo (N=60)
small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
elective surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — patient was hospitalized for elective total knee replacement
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin (N=58) | Placebo (N=60)
blurry eyes (Eye disorders) | 2 | 0
dry eyes (Eye disorders) | 4 | 0
constipation (Gastrointestinal disorders) | 2 | 1
dry mouth (Gastrointestinal disorders) | 4 | 2
diarrhea (Gastrointestinal disorders) | 2 | 4
upset stomach (Gastrointestinal disorders) | 3 | 1
nausea (Gastrointestinal disorders) | 3 | 2
vomiting (Gastrointestinal disorders) | 4 | 1
cold (Infections and infestations) | 9 | 4
pneumonia (Infections and infestations) | 2 | 0
UTI (Infections and infestations) | 2 | 1
headache (Nervous system disorders) | 2 | 3
worsening incontinence (Renal and urinary disorders) | 0 | 3
increased urinary frequency (Renal and urinary disorders) | 3 | 1
hot flashes (Reproductive system and breast disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No